CLINICAL TRIAL: NCT03932084
Title: Effects of Glucose Fluctuation Intervention on the Prognosis of Patients With Type 2 Diabetes and Cerebral Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Lou Qingqing, Director of Health Education Department, Nanjing University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N2017003
Record Dates: First submitted 2019-04-23; First posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Type 2 Diabetes and Cerebral Infarction
Keywords: Type 2 diabetes; Cerebral infarction; Glucose fluctuation targeted intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cerebral Infarction | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): During hospitalization:
  1. Monitor subjects' blood glucose;
  2. One-on-one education: Education includes skills related to diabetes self-management, basic knowledge of diabetes, diet, exercise, medication, blood glucose monitoring, risks of glucose fluctuations;
  3. Teaching patients and their families to use blood glucose meters and correctly record results. The diabetes specialist nurses demonstrate correct methods for self-monitoring blood glucose.
  During discharge: Patients were given standard hospital discharge instructions and were asked to monitor their blood glucose 5 times daily after discharge.
  Follow-up: If a patient FPG was less than 7 mmol/L, 2hPG was less than 10 mmol/L, or A1c was less than 7%, no intervention would be implemented. If one of these items was above the numbers, a referral would be made to an endocrinologist for medication adjustment. Participants received telephone follow-up one week after discharge, thereafter, follow-up were conducted once a month.
  Interventions: Behavioral: Control group
- Glucose fluctuation targeted intervention (Experimental): We set achieving goals for this intervention group (both A1c<7% and LAGE<80mg/dl). Participants received the same usual care as the control group; though additional attention was paid to glucose fluctuation on the basis of glucose control. Even the patient's FPG, 2hPG, and A1c were all well controlled, If his or her LAGE≥80mg/dl, we would carefully assess the patient's diet and exercise and daily activities first. If it was caused by lifestyle or events, the researchers worked with patients to find a self-care behavioral solution for the glucose fluctuation, and set behavioral goals, otherwise, the researchers would refer the patient to an endocrinologist for medication adjustment. During next follow-up, we evaluated the glucose fluctuation and target completion.
  Interventions: Behavioral: Glucose fluctuation targeted intervention

INTERVENTIONS:
Behavioral: Control group — During hospitalization:
  1. Monitor subjects' blood glucose;
  2. One-on-one education: Education includes skills related to diabetes self-management, basic knowledge of diabetes, diet, exercise, medication, blood glucose monitoring, risks of glucose fluctuations;
  3. Teaching patients and their families to use blood glucose meters and correctly record results. The diabetes specialist nurses demonstrate correct methods for self-monitoring blood glucose.
  During discharge: Patients were given standard hospital discharge instructions and were asked to monitor their blood glucose 5 times daily after discharge.
  Follow-up: If a patient FPG was less than 7 mmol/L, 2hPG was less than 10 mmol/L, or A1c was less than 7%, no intervention would be implemented. If one of these items was above the numbers, a referral would be made to an endocrinologist for medication adjustment. Participants received telephone follow-up one week after discharge, thereafter, follow-up were conducted once a month.
  Arms: Control group
Behavioral: Glucose fluctuation targeted intervention — We set achieving goals for this intervention group (both A1c<7% and LAGE<80mg/dl). Participants received the same usual care as the control group; though additional attention was paid to glucose fluctuation on the basis of glucose control. Even the patient's FPG, 2hPG, and A1c were all well controlled, If his or her LAGE≥80mg/dl, we would carefully assess the patient's diet and exercise and daily activities first. If it was caused by lifestyle or events, the researchers worked with patients to find a self-care behavioral solution for the glucose fluctuation, and set behavioral goals, otherwise, the researchers would refer the patient to an endocrinologist for medication adjustment. During next follow-up, we evaluated the glucose fluctuation and target completion.
  Arms: Glucose fluctuation targeted intervention

SUMMARY:
The present randomized control trial sought to establish glucose fluctuation as an important target for management on metabolic index, neurologic function, and quality of life in Type 2 diabetes mellitus (T2DM) patients and cerebral infarction (CI).

DETAILED DESCRIPTION:
There is a significant association between glycemic ﬂuctuation and the incidence of diabetes macrovascular complications. Therefore, understanding the impact of glycemic fluctuations on diabetic macroangiopathy could be helpful for discovering a strategy of prevention and treatment of macroangiopathy in diabetes. However, previous studies on the glycemic fluctuation in T2DM patients with CI were cross-sectional studies, there has been no prospective intervention study confirming the effects of glucose fluctuation targeted management on the prognosis of T2DM patients following CI. Based on previous fingdings, investigators will assess the effects of glucose fluctuation targeted intervention on metabolic index, neurologic function, and quality of life in T2DM patients and CI.

ELIGIBILITY:
Inclusion Criteria:

* 1. cerebral infarction within one month, diagnosed by magnetic resonance imaging (MRI) or computed tomography (CT) according to 1995 acute cerebral infarction diagnosis standards promulgated by the Fourth National Cerebrovascular Disease Conference [1];
* 2. having type 2 diabetes mellitus (as defined by the WHO diagnostic criteria in 1999) [2];

Exclusion Criteria:

* 1. coexisting acute complications of diabetes including diabetic ketoacidosis (DKA), hyperglycemic hyperosmolar syndrome (HHS), metabolic acidosis;
* 2. severe comorbid chronic complications of diabetes;
* 3. active malignancy;
* 4. subjects with mental illness and communication disorders; 5) those actively participating in other research studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-05-25 (Estimated); Study Completion 2019-06-18 (Estimated)

PRIMARY OUTCOMES:
Stroke severity | 6 months
  The National Institute of Health Stroke Scale includes the following domains: level of consciousness, sensory, neglect, visual field, gaze, facial palsy, motor arm, motor leg, limb ataxia, language, and dysarthria. Each domain is scored on an ordinal scale ranging from 0 to 2, 0 to 3, or 0 to 4. Item scores are summed to a total score ranging from 0 to 42 (the higher the score, the more severe the stroke).
Glycemic variability | 6 months
  fasting plasma glucose variation coefficient (CV-FPG)
Glucose fluctuation | 6 months
  Largest amplitude of Glycemic Excursions (LAGE)

SECONDARY OUTCOMES:
Disability and health-related quality of life after stroke | 6 months
  The Stroke Impact Scale (SIS) is a specific scale that evaluates disability and health-related quality of life after stroke. This scale includes the following eight domains: strength, memory, thinking, emotion, communication and ADLs, mobility, hand function and participation. A total of 8 domains with 59 items, are scored on a 5-point scale, of which the sixth, eighth, and ninth questions of the emotional dimension are reversed, and the other items are positive. Each domain scores range from 0 to 100 and are calculated using the following equation: Calculated score=[(actual score- the lowest possible score in this domain) / (the difference between the highest possible score and the lowest score in this domain)]×100. The total score of the scale is the sum of all domains. A higher score indicates better quality of life and the less functional damage.
Independent living skills | 6 months
  The Modified Rankin Scale can discriminate clinically relevant levels of disability and recovery in clinical trials. The 0-6 Likert scale is as follows: 0-no symptoms; 1-no significant disability; 2-slight disability; 3-moderate disability; 4-moderately severe disability; 5-severe disability; and 6-dead. The higher the score, the worse the patient's prognosis. When evaluating prognosis, a score≦2 was classified as a "good".
Glycemic control | 6 months
  Fasting plasma glucose (FPG), 2 hours postprandial blood glucose (2hPG), hemoglobin A1c (HbA1c) will be measured at 6 months.
Blood lipids | 6 months
  High-density lipoprotein-cholesterol (HDL-c), low-density lipoprotein-cholesterol (LDL-c), total cholesterol (TC), triglycerides (TG) will be measured at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Qingqing Lou, director, Principal Investigator — Nanjing University of Traditional Chinese Medicine
Locations (1):
- Affiliated Hospital of Integrated Traditional Chinese and Western Medicine, Nanjing University of Chinese Medicine, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Wu CH, Liu B. The Fourth National Cerebrovascular Disease Conference. China Medical News (6): 4, 1996.
- [Background] Colman PG, Thomas DW, Zimmet PZ, Welborn TA, Garcia-Webb P, Moore MP. New classification and criteria for diagnosis of diabetes mellitus. The Australasian Working Party on Diagnostic Criteria for Diabetes Mellitus. N Z Med J. 1999 Apr 23;112(1086):139-41. PMID 10340693
- [Derived] Lou Q, Yuan X, Hao S, Miller JD, Yan J, Zuo P, Li J, Yang L, Li H. Effects of Glucose Fluctuation Targeted Intervention on the Prognosis of Patients with Type 2 Diabetes following the First Episode of Cerebral Infarction. J Diabetes Res. 2020 Jan 28;2020:2532171. doi: 10.1155/2020/2532171. eCollection 2020. PMID 32090117